CLINICAL TRIAL: NCT00395395
Title: A Partially-Blind, Randomized, Single-Dose, Placebo-Controlled Crossover Phase I Study Assessing the Effect of Water and Food Intake on the Pharmacokinetics and Pharmacodynamics of SMC021 0.8 mg in Healthy Postmenopausal Women
Brief Title: Effects of Water and Food Intake on the Pharmacokinetics and Pharmacodynamics of Oral Salmon Calcitonin in Healthy Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CSMC021A2112
Record Dates: First submitted 2006-10-31; First posted 2006-11-02 (Estimated); Last update posted 2007-05-28 (Estimated); Status verified 2007-05

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Postmenopausal; osteoporosis; Pharmacokinetics/dynamics; Calcitonin
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — salmon calcitonin

INTERVENTIONS:
Drug: Oral salmon calcitonin, salmon calcitonin nasal spray

SUMMARY:
This is a phase I study to analyze the effect of water and food intake on the bioavailability and pharmacodynamic of oral salmon calcitonin (SMC021) and salmon calcitonin nasal spray in post-menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal women

Exclusion Criteria:

* Previous treatment with other osteoporosis medication

Other protocol defined inclusion/exclusion criteria may apply.

Ages: 40 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2006-10

PRIMARY OUTCOMES:
Pharmacokinetic (PK) profile of oral salmon calcitonin taken in the morning with 50 ml or 200 ml water and at 10, 30 or 60 minutes before a meal

SECONDARY OUTCOMES:
Pharmacodynamic (PD) profile of oral salmon calcitonin taken in the morning with 50 ml or 200 ml water and at 10, 30 or 60 minutes before a meal
PK profile of the carrier of oral salmon calcitonin, taken in the morning with 50 ml or 200 ml water and at 10, 30 or 60 minutes before a meal
PK profile of salmon calcitonin nasal spray

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Basel, Study Director — Novartis Basel +41 61 324 1111
Locations (1):
- Multiple Cities, Denmark